CLINICAL TRIAL: NCT02875470
Title: Diamond Burs Versus Gracey Curettes and Efficacy of Root Planing in Chronic Periodontitis Patients
Brief Title: Burs Versus Curettes in Root Planing.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Principal Investigator, Fatma Türktekin, Principal investigator, Ege University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FTurktekin
Record Dates: First submitted 2016-08-09; First posted 2016-08-23 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Periodontitis
Keywords: non-surgical periodontal debridement; root planing/instrumentation; cytokine(s); dental plaque; microscopy, electron, scanning
MeSH Terms: conditions — Chronic Periodontitis; Dental Plaque

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensiv Perio Set (Experimental): Root planing with diamond burs
  Interventions: Device: Intensiv Perio Set
- Gracey curette (Active Comparator): Root planing with Gracey curettes
  Interventions: Device: Gracey curette

INTERVENTIONS:
Device: Intensiv Perio Set — Diamond burs for root planing
  Arms: Intensiv Perio Set
Device: Gracey curette
  Arms: Gracey curette

SUMMARY:
This study compares the efficacy of diamond burs and Gracey curettes in non-surgical periodontal treatment of chronic periodontitis by clinical, microbiological, biochemical parameters and scanning electron microscopic investigations on root surfaces. Two quadrants of each of the 12 patients were treated with diamond burs whereas other 2 quadrants were treated with Gracey curettes. Also 21 hopeless teeth received root planing either with diamond burs or curettes or no treatment at all and were then extracted for microscopic evaluations.

DETAILED DESCRIPTION:
Gracey curettes are the most widely used instruments for root planing and regarded as the gold standard, but their usage is technic sensitive and time consuming for the clinician and efficacy reduces in deep pockets, root irregularities, and furcations. Alternative sonic, ultrasonic and rotary instruments have been investigated for potential benefits in improving mechanical access. Sonic and ultrasonic instruments are used for scaling, but they cannot provide smooth root surfaces.

Intensiv Perio Set is a rotating diamond bur system developed for odontoplasty, scaling and root planing. It is used only in right angle hand piece, at rotation speeds of 6000 rpm, with reduced pressure application. These burs have two different head types for morphologically different areas; flame or tapered, three different grains; 75, 40, or 15 μm, with either a short or long neck for each unit. Burs with 75 μm grain are used only in odontoplasty, whereas, 40 and 15 μm burs are used for scaling and root planing.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of generalized chronic periodontitis (Armitage 1999)
* presence of at least 3 teeth (1 molar, 2 non-molar teeth) with probing depth ≥ 5 mm in each quadrant

Exclusion Criteria:

* presence of any known systemic disease or using medications that affect periodontal tissues
* antibiotic treatment and/or periodontal treatment within the past 6 months
* tobacco usage during the last 12 months
* being pregnant or in the lactation period

Ages: 37 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Clinical tissue healing | 6 month

SECONDARY OUTCOMES:
Changing of the amount of pathogen microorganisms | 1 month
Changing of the gingival crevicular fluid biomarkers | 1 month
Root surface characteristic according to Scanning Electron Microscope | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Eralp Buduneli, Proffessor, Study Director — Department of Periodontology, Faculty of Dentistry, Ege University

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data for all outcome measures will be made available within 3 years of study completion.